CLINICAL TRIAL: NCT02715973
Title: Nutritional Assessment Tool and Nutritional Intervention in Childhood Chronic Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-CLD-Nutrition-01
Record Dates: First submitted 2016-02-17; First posted 2016-03-22 (Estimated); Last update posted 2018-12-06 (Actual); Status verified 2017-12

CONDITIONS: Chronic Liver Disease
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nutritional Supplement (Experimental): Diet Counseling (Energy=200 kcal/kg/day, (present weight) protein =3-4 gm/kg/day)
  Nutritional supplement (Providing extra 40 kcal/kg/day)
  Interventions: Dietary Supplement: Nutritional Supplement
- Standard nutritional treatment (Active Comparator): Diet counselling only (Energy=200 kcal/kg/day (present weight) protein =3-4 gm/kg/day).
  Standard nutritional treatment
  Interventions: Dietary Supplement: Standard Nutritional Treatment

INTERVENTIONS:
Dietary Supplement: Nutritional Supplement — Energy dense supplement appox. 2 kcal/mL, prepared from locally available, affordable, socially acceptable food items - milk, sugar, edible coconut oil, egg and custard powder as base) in addition to standard nutritional counseling by a trained dietician as per the recommended daily allowance according to gender and age.
  Arms: Nutritional Supplement
Dietary Supplement: Standard Nutritional Treatment — Standard nutritional counseling by a trained dietician as per the recommended daily allowance according to gender and age
  Arms: Standard nutritional treatment

SUMMARY:
Children (Exclusively breast fed: 6mo - 3yrs, and who are not exclusively breast fed 3mo to 3 yrs) with infantile cholestasis syndrome will be randomized to either recieve indigenously prepared oral nutritional supplement (energy dense supplement appox. 2 kcal/mL, prepared from locally available, affordable, socially acceptable food items - milk, sugar, edible coconut oil, egg and custard powder as base) in addition to standard nutritional counseling by a trained dietician (Group A). The control group (Group B) in comparison will receive standard nutritional counseling from a trained dietician but will not receive any additional nutritional supplement. All the children will be followed up at 1 month, 3 months, 6 months, 9 months and 1 year after inclusion. Clinical, nutritional assessment and laboratory data will be collected at each visit. Additionally IL-6 levels will be done at each visit in children of both arms of the intervention group.

The outcomes of interest will be growth and improvement of nutritional status parameters, hepatic morbidity (ascites, gastrointestinal bleeding, encephalopathy, {SBP (Spontaneous Bacterial Peritonitis), HRS (Hepatorenal Syndrome), etc and outcome (improvement, death or Liver Transplantation}.

All children will receive individualized standard treatment for infantile cholestasis syndrome including vitamin supplements/endotherapy/ beta blockers/ prophylaxis for SBP (Spontaneous Bacterial Peritonitis)/cholangitis (to at risk children) and drug therapy wherever indicated (steroids/ copper chelation/ UDCA).

ELIGIBILITY:
Inclusion Criteria:

1. Nutritional intervention in children with moderate and severe malnutrition as pr standard anthropometric measures children (Exclusively breast fed: 6mo - 3yrs, and who are not exclusively breast fed : 3mo to 3 yrs) with infantile cholestasis syndrome)
2. Hindi/English speaking family

Exclusion Criteria:

1. Any metabolic or endocrinal diseases independently affecting nutritional status
2. Refusal to give written informed consent to participate in the study

Ages: 3 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
To study the effect of special fortified indigenous diet on growth,and outcome in children with infantile cholestasis syndrome | 1 year
  Growth is a composite outcome defines as age and sex appropriate anthropometric measures- weight , height, mid arm circumference, triceps skin fold thickness, subscapular skin fold thickness.
To study the effect of special fortified indigenous diet on hepatic morbidity in children with infantile cholestasis syndrome | 1 year
  hepatic morbidity is a composite outcome comprising of ascites, hepatic encephalopathy, spontaneous bacterial peritonitis, intercurrent infections, variceal bleed.
To study the effect of special fortified indigenous diet on outcome in children with infantile cholestasis syndrome | 1 year
  Outcome is defined as survival with native liver, death or liver transplantation

SECONDARY OUTCOMES:
To study the levels of IL-6 before & after nutritional therapy in malnourished children with Chronic Liver Disease | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dr Seema Alam, MD, Study Director — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided